CLINICAL TRIAL: NCT05601076
Title: Design and Application of Small-diameter Closed Thoracic Drainage Tube Fixation Following Lung Wedge Resection: a Randomised Prospective Study
Brief Title: Small-diameter Closed Thoracic Drainage Tube Fixation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Caifang Yang, director, Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Taizhouhospital002
Record Dates: First submitted 2022-10-20; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Wedge Resection

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The drainage tube in the experimental group was fixed with the triple-buffer system (Experimental)
  Interventions: Procedure: fixed with the triple-buffer system
- that in the control group was fixed using the conventional lifting platform method (Active Comparator)
  Interventions: Procedure: fixed using the conventional lifting platform method

INTERVENTIONS:
Procedure: fixed with the triple-buffer system — The steps were as follows: i) elastic cotton tape (3M 2733-25 Japan Ltd., Tokyo, Japan) was used at the proximal 15 cm from the incision, with 5 × 2.5 cm pieces glued to the skin and fixed with the drainage tube using surgical knots; ii) the distal end of the ligation was fixed using the same method, while the ligation position was higher than the first; iii) the ligature point was fixed next to the elastic soft cotton tape (5 × 5 cm), using the high-platform method to fix the drainage tube, with the drainage tube curved; and iv) the drainage tube between the two fixed points was inserted with a specific radian.
  Arms: The drainage tube in the experimental group was fixed with the triple-buffer system
Procedure: fixed using the conventional lifting platform method — In terms of the control group, two lines of flexible cotton tape (3M 2733-25 Japan Ltd., Tokyo, Japan) measuring 10 × 2.5 cm were used, and the drainage tube was fixed parallel to the long axis and glued to the middle-position 360° winding tube once the drainage tube was 0.5 cm higher than the surrounding skin. Next, the drainage tube was fixed at both ends to the patient's skin using adhesive tape. Then, the tube and the adhesive plaster were overlapped vertically and horizontally, the tube was inserted, the adhesive plaster was added, and then the chest tube was fixed on the adhesive plaster by knotting the interspersed cotton rope, which was equal to indirectly fixing the tube on the patient's skin
  Arms: that in the control group was fixed using the conventional lifting platform method

SUMMARY:
Objective: To explore the design feasibility and application effect of triple-buffer-system-fixed small-diameter (18 F) thoracic closed drainage tubes following lung wedge resection. Methods: A total of 136 patients with indwelling thoracic drainage tubes following pulmonary wedge resection were recruited, with 70 patients allocated to the control group and 66 to the experimental group. The drainage tube in the experimental group was fixed with the triple-buffer system, while that in the control group was fixed using the conventional lifting platform method. The incidence of unplanned extubation, the indwelling time of the drainage tube and the time and material costs, as well as information regarding any subcutaneous emphysema and skin tension blisters, were recorded following the operation. The pain and degree of comfort were assessed using a chi-square test and a rank sum t-test to compare the differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Single-port thoracoscopic wedge resection of the lung was performed for the first time
* No air leak in the lung tissue was detected
* The patient could communicate and cooperate normally.
* No local skin allergy or scar could be observed.

Exclusion Criteria:

* Patients with wide adhesion of the whole thoracic mucosa.
* Patients with postoperative or intraoperative bleeding.
* Patients with severe postoperative hypoproteinaemia or chylothorax with massive pleural effusion.
* Patients diagnosed with emphysema.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The extubation standard | 2 hours
  The extubation standard is patients with good lung re-expansion after clamping for 24 h and no obvious air leakage after reopening the chest tube, and a drainage volume of <250 mL within 24 h, which can be removed.
the pain numerical rating scale | 2 hours
  no pain: 0 points, mild pain: 1-3 points, moderate pain: 4-7 points and severe pain: 8-10 points
the Kolcaba comfort scalea(four-point scale) | 2 hours
  1: strongly disagree, 2: disagree, 3: agree, 4: strongly agree
The adverse reactions | 2 hours
  The chest skin was bulged, and the gas could be felt in the subcutaneous tissue through hand pressing, and there was a feeling of twisting or snow grip.

CONTACTS AND LOCATIONS:
Overall Officials: Caifang Yang, Dr., Study Director — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou, Zhejiang, China